CLINICAL TRIAL: NCT00333359
Title: An Open-Label, 52-Week Extension Study Assessing XP13512 Safety and Efficacy in Patients With Restless Legs Syndrome.
Brief Title: XP13512 (Gabapentin Enacarbil) Extension Study in Patients With Restless Legs Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111490
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XP13512 (GEn) (Experimental): 1200 mg XP13512, orally, once daily for 52 weeks
  Interventions: Drug: XP13512 (GEn)

INTERVENTIONS:
Drug: XP13512 (GEn) — 1200 mg XP13512, orally, once daily for 52 weeks
  Other Names: GSK1838262; Gabapentin Enacarbil

SUMMARY:
The primary objective of this trial is to assess the long-term safety and efficacy of XP13512 (Gabapentin Enacarbil) taken once daily for the treatment of patients suffering from Restless Legs Syndrome (RLS).

DETAILED DESCRIPTION:
Study XP055 is a multicenter, open-label, 52-week extension study of XP13512 (Gabapentin Enacarbil [GEn]) given once daily to eligible subjects with Restless Legs Syndrome (RLS) who had previously completed 1 of the following studies and met eligibility criteria: XP052 (110963 [NCT00298623]), XP053 (111460 [NCT00365352]), XP081 (111462 [NCT01332305]), and XP083 (111463 [NCT01332318]).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed one of the following studies: XP052 (110963 [NCT00298623]), XP053 (111460 [NCT00365352]), XP081 (111462 [NCT01332305]), and XP083 (111463 [NCT01332318]).

Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, would be non-compliant with the study visit schedule, procedures, or medication administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Ellenbogen AL, Thein SG, Winslow DH, Becker PM, Tolson JM, Lassauzet ML, Chen D. A 52-week study of gabapentin enacarbil in restless legs syndrome. Clin Neuropharmacol. 2011 Jan-Feb;34(1):8-16. doi: 10.1097/WNF.0b013e3182087d48. PMID 21242741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants completing one of four parent studies (110963 [NCT00298623], 111460 [NCT00365352], 111462 [NCT01332305], and 111463 [NCT01332318]) were eligible to enroll in Study 111490 (NCT00333359) if eligibility criteria were met.
Groups:
- Naïve; 1200 mg GEn: Naïve participants received placebo (therefore naïve to gabapentin enacarbil [GEn]) in a parent study, followed by GEn 1200 mg once a day (with the flexibility to go up to 1800 mg or down to 600 mg based on tolerability and efficacy) in this study.
- Non-naïve; 1200 mg GEn: Non-naïve participants received GEn in a parent study, followed by GEn 1200 mg once a day (with the flexibility to go up to 1800 mg or down to 600 mg based on tolerability and efficacy) in this study.
Period: Overall Study
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn
Started | 199 | 382
Completed | 126 | 260
Not Completed | 73 | 122
Not completed — Adverse Event | 29 | 35
Not completed — Withdrawal by Subject | 19 | 37
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Non-compliance | 2 | 8
Not completed — Lost to Follow-up | 15 | 25
Not completed — Termination or Withdrawal by Sponsor | 1 | 1
Not completed — Treatment Failure | 3 | 8
Not completed — Withdrew before Receiving One Dose | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | Total
Number analyzed (Participants) | 197 | 376 | 573
Age Continuous [Mean (Standard Deviation); unit: Years] — The Safety Population, consisting of all participants who were enrolled in the study and took at least 1 dose (or any portion of a dose) of study medication, was used for summarizing all baseline characteristics. Eight enrolled participants did not meet the criteria for inclusion in the Safety Population.
  Years | 49.5 (12.03) | 50.6 (11.82) | 50.2 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants] — The Safety Population, consisting of all participants who were enrolled in the study and took at least 1 dose (or any portion of a dose) of study medication, was used for summarizing all baseline characteristics. Eight enrolled participants did not meet the criteria for inclusion in the Safety Population.
  Participants
    Female | 119 | 217 | 336
    Male | 78 | 159 | 237
Race/Ethnicity, Customized [Number; unit: participants] — The Safety Population, consisting of all participants who were enrolled in the study and took at least 1 dose (or any portion of a dose) of study medication, was used for summarizing all baseline characteristics. Eight enrolled participants did not meet the criteria for inclusion in the Safety Population.
  participants
    White or Caucasian | 192 | 360 | 552
    American Indian or Alaskan Native | 1 | 5 | 6
    Asian | 1 | 3 | 4
    Black or African American | 2 | 5 | 7
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Unknown | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the International Restless Legs Syndrome Rating Scale (IRLS) at Week 52 Using Observed Case (OC)
Description: The IRLS rating scale is a measure of RLS disease severity. The score reflects participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Also, items are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total score on the IRLS ranges from 0 to 40, with higher values representing more severe RLS symptoms. Change from baseline was calculated as the Week 52 value minus the baseline value. Change scores with higher value represents greater improvement in RLS symptoms.
Time Frame: Baseline and Week 52
Population: Safety Population: all participants who received one dose or any part of one dose of GEn. Week 52 (end of treatment) results included only Week 52 observed cases and do not include early termination values; as such, the number of participants analyzed differs from the number of participants in the Baseline Characteristics summary.
Measure: Mean (Standard Deviation); unit: points on a scale
Groups:
- All Participants; 1200 mg GEn: All participants received GEn or placebo in a parent study, followed by GEn 1200 mg once a day (with the flexibility to go up to 1800 mg or down to 600 mg based on tolerability and efficacy) in this study.
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 125 | 254 | 379
points on a scale | -16.3 (8.23) | -17.0 (8.20) | -16.8 (8.21)

2. Primary Outcome: Number of Participants Classified as Responders to Treatment on the Investigator-rated Clinical Global Impressions of Improvement (CGI-I) at Each Visit Using OC
Description: The CGI-I is a widely used tool designed to allow clinicians to rate the severity of illness and the change over time based on a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to the start of the study. Responders on the CGI-I are defined as those with a score of 1 or 2, corresponding to "very much improved" or "improved," respectively.
Time Frame: Weeks 0, 1, 4, 12, 24, 36, and 52
Population: Safety Population. Results at each week include only observed cases and do not include early termination values; as such, the number of participants analyzed differs from the number of participants in the Baseline Characteristics summary.
Measure: Number; unit: participants
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 197 | 376 | 573
participants
  Week 0, n=197, 376, 573 | 84 | 300 | 384
  Week 1, n=185, 363, 548 | 152 | 294 | 446
  Week 4, n=171, 354, 525 | 143 | 308 | 451
  Week 12, n=150, 324, 474 | 133 | 297 | 430
  Week 24, n=138, 305, 443 | 126 | 275 | 401
  Week 36, n=132, 281, 413 | 120 | 260 | 380
  Week 52, n=126, 262, 388 | 115 | 247 | 362

3. Secondary Outcome: Change From Baseline in the IRLS Rating Scale Score at Each Visit Using OC
Description: The IRLS rating scale is a measure of RLS disease severity. The score reflects participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Also, items are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total score on the IRLS ranges from 0 to 40, with higher values representing more severe RLS symptoms. Change from baseline was calculated as the value at each visit minus the baseline value. Change scores with higher values represent greater improvement in RLS symptoms.
Time Frame: Weeks 0, 1, 4, 12, 24, and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 197 | 376 | 573
points on a scale
  Week 0, n=197, 376, 573 | -9.4 (8.08) | -14.6 (8.40) | -12.8 (8.64)
  Week 1, n=186, 360, 546 | -15.6 (7.44) | -13.5 (8.47) | -14.2 (8.19)
  Week 4, n=174, 352, 526 | -15.6 (7.72) | -15.8 (7.80) | -15.7 (7.77)
  Week 12, n=150, 322, 472 | -15.8 (8.76) | -16.3 (7.84) | -16.1 (8.14)
  Week 24, n=139, 305, 444 | -16.2 (7.53) | -16.5 (7.80) | -16.4 (7.71)
  Week 36, n=130, 281, 411 | -16.8 (7.79) | -16.6 (8.23) | -16.7 (8.09)

4. Secondary Outcome: Number of Participants in Each Category of the Investigator-rated CGI-I by Visit Using OC
Description: The CGI-I is a widely used tool designed to allow clinicians to rate the severity of illness and the change over time based on a seven-point rating scale, with a score of 1 being "very much improved," 2 being "much improved," 3 being "minimally improved," 4 being "no change," 5 being "minimally worse," 6 being "much worse," and 7 being "very much worse" compared to the start of the study.
Time Frame: Weeks 0, 1, and 52
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 197 | 376 | 573
participants
  Week 0, Very much improved, n=197, 376, 573 | 38 | 192 | 230
  Week 0, Much improved, n=197, 376, 573 | 46 | 108 | 154
  Week 0, Minimally improved, n=197, 376, 573 | 47 | 37 | 84
  Week 0, No change, n=197, 376, 573 | 55 | 36 | 91
  Week 0, Minimally worse, n=197, 376, 573 | 9 | 0 | 9
  Week 0, Much worse, n=197, 376, 573 | 2 | 2 | 4
  Week 0, Very much worse, n=197, 376, 573 | 0 | 1 | 1
  Week 1, Very much improved, n=185, 363, 548 | 82 | 155 | 237
  Week 1, Much improved, n=185, 363, 548 | 70 | 139 | 209
  Week 1, Minimally improved, n=185, 363, 548 | 28 | 40 | 68
  Week 1, No change, n=185, 363, 548 | 4 | 25 | 29
  Week 1, Minimally worse, n=185, 363, 548 | 0 | 3 | 3
  Week 1, Much worse, n=185, 363, 548 | 1 | 1 | 2
  Week 1, Very much worse, n=185, 363, 548 | 0 | 0 | 0
  Week 52, Very much improved, n=126, 262, 388 | 72 | 187 | 259
  Week 52, Much improved, n=126, 262, 388 | 43 | 60 | 103
  Week 52, Minimally improved, n=126, 262, 388 | 7 | 9 | 16
  Week 52, No change, n=126, 262, 388 | 4 | 4 | 8
  Week 52, Minimally worse, n=126, 262, 388 | 0 | 0 | 0
  Week 52, Much worse, n=126, 262, 388 | 0 | 1 | 1
  Week 52, Very much worse, n=126, 262, 388 | 0 | 1 | 1

5. Secondary Outcome: Number of Participants Classified as Responders to Treatment on the Participant-rated CGI-I at Each Visit Using OC
Description: The Participant-rated CGI-I is a self-reported measure completed by the participant, who rates the change from the start of the study in the severity of their illness using a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse". Responders on the Participant-rated CGI-I are defined as those with a score of 1 or 2, corresponding to "very much improved" and "improved," respectively.
Time Frame: Weeks 0, 1, 4, 12, 24, 36, and 52
Population: Safety Population. Results at each week include only observed cases and do not include early termination values; as such, the number of participants analyzed at each week differs from the number of participants in the Baseline Characteristics summary.
Measure: Number; unit: participants
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 197 | 376 | 573
participants
  Week 0, n=197, 376, 573 | 86 | 304 | 390
  Week 1, n=182, 351, 533 | 145 | 261 | 406
  Week 4, n=171, 348, 519 | 143 | 299 | 442
  Week 12, n=148, 318, 466 | 131 | 283 | 414
  Week 24, n=133, 300, 433 | 117 | 275 | 392
  Week 36, n=129, 276, 405 | 115 | 252 | 367
  Week 52, n=122, 247, 369 | 107 | 227 | 334

6. Secondary Outcome: Number of Participants in Each Category of the Participant-rated CGI-I by Visit Using OC
Description: The Participant-rated CGI-I is a self-reported measure completed by the participant who rates the change from the start of the study in the severity of their illness using a seven-point rating scale, with a score of 1 being "very much improved," 2 being "much improved," 3 being "minimally improved," 4 being "no change," 5 being "minimally worse," 6 being "much worse," and 7 being "very much worse" compared to the start of the study.
Time Frame: Weeks 0, 1, and 52
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 197 | 376 | 573
participants
  Week 0, Very much improved, n=197, 376, 573 | 39 | 194 | 233
  Week 0, Much improved, n=197, 376, 573 | 47 | 110 | 157
  Week 0, Minimally improved, =197, 376, 573 | 47 | 35 | 82
  Week 0, No change, n=197, 376, 573 | 50 | 29 | 79
  Week 0, Minimally worse, n=197, 376, 573 | 8 | 6 | 14
  Week 0, Much worse, n=197, 376, 573 | 5 | 1 | 6
  Week 0, Very much worse, n=197, 376, 573 | 1 | 1 | 2
  Week 1, Very much improved, n=182, 351, 533 | 91 | 171 | 262
  Week 1, Much improved, n=182, 351, 533 | 54 | 90 | 144
  Week 1, Minimally improved, n=182, 351, 533 | 29 | 48 | 77
  Week 1, No change, n=182, 351, 533 | 4 | 28 | 32
  Week 1, Minimally worse, n=182, 351, 533 | 1 | 6 | 7
  Week 1, Much worse, n=182, 351, 533 | 2 | 7 | 9
  Week 1, Very much worse, n=182, 351, 533 | 1 | 1 | 2
  Week 52, Very much improved, n=122, 247, 369 | 80 | 177 | 257
  Week 52, Much improved, n=122, 247, 369 | 27 | 50 | 77
  Week 52, Minimally improved, n=122, 247, 369 | 11 | 13 | 24
  Week 52, No change, n=122, 247, 369 | 3 | 5 | 8
  Week 52, Minimally worse, n=122, 247, 369 | 0 | 0 | 0
  Week 52, Much worse, n=122, 247, 369 | 0 | 1 | 1
  Week 52, Very much worse, n=122, 247, 369 | 1 | 1 | 2

7. Secondary Outcome: Number of Participants With no Reported RLS Symptoms During Each of the 4-hour Periods From the 24-hour RLS Record at Week 52 Using OC Data
Description: In the 24-Hour RLS Record (diary), participants report the presence and severity of RLS symptoms (none, mild, moderate, or severe) for a 24-hour period, in 30-minute increments. The period was divided into 7 four-hour intervals (8 AM to 12PM, 12 to 4PM, 4 to 8PM, 6 to 10PM, 8 to 12 Midnight, Midnight to 4AM, 4 to 8AM).
Time Frame: Week 52
Population: Safety Population. Results at Week 52 include only Week 52 observed cases and do not include early termination values; as such, the number of participants with data at each time point differs from the number of participants in the Baseline Characteristics summary.
Measure: Number; unit: participants
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 123 | 241 | 364
participants
  8 AM to 12 PM, n=123, 241, 364 | 106 | 224 | 330
  12 PM to 4 PM, n=122, 240, 362 | 106 | 216 | 322
  4 PM to 8 PM, n=122, 240, 362 | 88 | 184 | 272
  6 PM to 10 PM, n=122, 241, 363 | 80 | 175 | 255
  8 PM to 12 AM, n=122, 241, 363 | 75 | 162 | 237
  12 AM to 4 AM, n=123, 241, 364 | 98 | 195 | 293
  4 AM to 8 AM, n=123, 241, 364 | 104 | 214 | 318

8. Secondary Outcome: Median Time to Onset of the First RLS Symptom Using the RLS Symptom Record at Weeks 24 and 52
Description: The 24-Hour RLS Record is a diary in which participants report the presence and severity of RLS symptoms for a 24-hour period, in 30-min increments, beginning at 8AM on the day prior to the visit.
Time Frame: Weeks 24 and 52
Population: Safety Population. Results include only observed cases and do not include early termination values; as such, the number of participants analyzed at each week differs from the number of participants in the Baseline Characteristics summary.
Measure: Median (Full Range); unit: hours
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 127 | 285 | 412
hours
  Week 24, n=127, 285, 412 | 15.5 [0 to 21] | 20 [0 to 24] | 18 [0 to 24]
  Week 52, n=123, 241, 364 | NA [0 to 19.5] — The median was not estimable with Kaplan-Meier methodology at Week 52 because fewer than 50% of participants experienced an event. | NA [0 to 19] — The median was not estimable with Kaplan-Meier methodology at Week 52 because fewer than 50% of participants experienced an event. | NA [0 to 19.5] — The median was not estimable with Kaplan-Meier methodology at Week 52 because fewer than 50% of participants experienced an event.

9. Secondary Outcome: Overall Quality of Life (QoL) Impact Score of the RLS Quality of Life Questionnaire at Weeks 24 and 52
Description: The RLS QoL is an 18-item scale assessing the impact of RLS on daily life, emotional well-being, social and work life. Responses range from 1 (not at all/never) to 5 (a lot/all of the time). Ten items contribute to a single summary score, the Overall Life Impact, which is standardized to range from 0-100, with lower scores representing better QoL.
Time Frame: Weeks 24 and 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 164 | 328 | 429
points on a scale
  Week 24, n=164, 328, 492 | 89.8 (12.27) | 91.1 (12.04) | 90.7 (12.12)
  Week 52, n=121, 264, 385 | 92.0 (9.77) | 92.0 (11.66) | 92.0 (11.09)

10. Secondary Outcome: Mean Change From Baseline at Week 24 and Week 52 in Work Productivity and Activity Impairment Questionnaire (WPAI:SHP) Summary Scores
Description: The WPAI:SHP estimates work productivity and social activities lost over the past week due to RLS symptoms. Each summary score is expressed as a percentage and ranges from 0 to 100, with higher scores indicating more work missed; a negative change from baseline indicates less work missed. Change = the observed value at the current visit minus the observed value at Week 0. Change is calculated only for participants who had a value at both the current visit and at Week 0.
Time Frame: Baseline and Weeks 24 and 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 158 | 309 | 467
percent change
  Week 24, Work Time Missed, n=108, 199, 307 | -0.2 (5.24) | 0.1 (4.88) | 0.0 (5.00)
  Week 24, Impairment While Working, n=101, 185, 286 | -7.6 (19.50) | -2.3 (10.80) | -4.2 (14.67)
  Week 24, Overall Work Impairment, n=101, 185, 286 | -7.6 (20.39) | -2.2 (11.80) | -4.1 (15.57)
  Week 24, Daily Activity Impairment, n=158,309,467 | -10.3 (20.11) | -4.3 (18.02) | -6.3 (18.95)
  Week 52, Work Time Missed, n=82, 175, 257 | -0.2 (7.16) | 1.0 (9.86) | 0.6 (9.09)
  Week 52, Impairment While Working n=78, 170, 248 | -8.7 (18.26) | -0.9 (5.61) | -3.3 (16.85)
  Week 52, Overall Work Impairment, n=78, 170, 248 | -8.9 (19.25) | -0.8 (17.03) | -3.3 (18.12)
  Week 52, Daily Activity Impairment, n=117,261,378 | -11.5 (20.31) | -3.9 (19.62) | -6.3 (20.11)

11. Secondary Outcome: Mean Change From Baseline at Week 24 and Week 52 in Work Productivity and Activity Impairment Questionnaire (WPAI:SHP) Individual Items: Hours of Work Missed Due to RLS, Hours of Work Missed Due to Other Reason, and Hours Actually Worked
Description: The WPAI:SHP estimates work productivity and social activities lost over the past week due to RLS symptoms. Change is calculated as the observed value at Week 24/52 minus the observed value at baseline. Absenteeism is recorded as the number of hours missed from work. W, Week; hr, hour.
Time Frame: Baseline and Weeks 24 and 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 108 | 199 | 307
hours
  W24, hr missed due to RLS, n=108, 199, 307 | -0.1 (1.08) | -0.1 (3.30) | -0.1 (2.73)
  W24, hr missed for other reason, n=108, 199, 307 | -1.8 (8.94) | -0.2 (12.56) | -0.8 (11.43)
  HW24, hr actually worked, n=108, 199, 307 | 0.8 (18.09) | 2.5 (17.60) | 1.9 (17.76)
  W52, hr missed due to RLS, n=82, 175, 257 | 0.1 (2.39) | 0.2 (4.10) | 0.2 (3.64)
  W52, hr missed other reason, n=82, 175, 257 | 0.5 (10.78) | -1.8 (11.58) | -1.0 (11.36)
  W52, hr actually worked, n=82, 175, 257 | 0.0 (19.79) | 2.2 (17.98) | 1.5 (18.56)

12. Secondary Outcome: Mean Change From Baseline at Weeks 24 and 52 in Work Productivity and Activity Impairment Questionnaire (WPAI:SHP) Individual Item: RLS Affected Productivity
Description: The WPAI:SHP estimates work productivity and social activities lost over the past week due to RLS symptoms. Change is calculated as the observed value at Week 52 minus the observed value at baseline. Productivity affected while working is estimated on a 0 (no effect) to 10 scale (completely preventing productivity).
Time Frame: Baseline and Weeks 24 and 52
Population: Safety Population: all participants who received one dose or any part of one dose of GEn. Results include only observed cases and do not include early termination values; as such the number of participants analyzed at each week differs from the number of participants in the Baseline characteristics summary.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Number analyzed (Participants) | 197 | 376 | 573
points on a scale
  Week 24, n=101, 185, 286 | -0.8 (1.95) | -0.2 (1.08) | -0.4 (1.47)
  Week 52, n=78, 170, 248 | -0.9 (1.83) | -0.1 (1.56) | -0.3 (1.68)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) and serious adverse event (SAE) collection started immediately following informed consent and continued throughout the study (up to Week 53).
Description: At the end of the follow-up period, Week 57 (30 days after the last day of taper), the study coordinator called participants to determine if any SAEs occurred, and the resolution date for any AEs that were ongoing at the end of the study.
Arm/Group | Naïve; 1200 mg GEn | Non-naïve; 1200 mg GEn | All Participants; 1200 mg GEn
Serious Adverse Events (participants affected / at risk) | 7/197 | 14/376 | 21/573
Other Adverse Events (participants affected / at risk) | 114/197 | 144/376 | 258/573
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naïve; 1200 mg GEn (N=197) | Non-naïve; 1200 mg GEn (N=376) | All Participants; 1200 mg GEn (N=573)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 (0) | 1
Herpes Zoster (Infections and infestations) | 1 | 0 (0) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 (0) | 1
Meningitis Viral (Infections and infestations) | 1 | 0 (0) | 1
Nerve Root Compression (Nervous system disorders) | 1 | 0 (0) | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 (0) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0) | 1
Angina Unstable (Cardiac disorders) | 0 (0) | 1 | 1
Appendicitis (Infections and infestations) | 0 (0) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 | 1
Chest Pain (General disorders) | 0 (0) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 (0) | 1 | 1
Drug Withdrawal Syndrome (General disorders) | 0 (0) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 | 1
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 | 1
Postoperative Infection (Infections and infestations) | 0 (0) | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naïve; 1200 mg GEn (N=197) | Non-naïve; 1200 mg GEn (N=376) | All Participants; 1200 mg GEn (N=573)
Somnolence (Nervous system disorders) | 54 | 59 | 113
Dizziness (Nervous system disorders) | 39 | 27 | 66
Headache (Nervous system disorders) | 15 | 26 | 41
Fatigue (General disorders) | 15 | 16 | 31
Nausea (Gastrointestinal disorders) | 10 | 20 | 30
Nasopharyngitis (Infections and infestations) | 8 | 20 | 28
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 15 | 25
Restless Legs Syndrome (Nervous system disorders) | 14 | 10 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.